CLINICAL TRIAL: NCT05894317
Title: Vascular Access Complications for Therapeutic Apheresis in Nephrology : a Retrospective Observational Study in North-East France.
Brief Title: Vascular Access Complications for Therapeutic Apheresis in Nephrology
Acronym: VACTANE
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, CORBEL Alice, Dr.CORBEL Alice Nephrology, MD, Central Hospital, Nancy, France
Other Study IDs: 2022PI162
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Vascular Access Complication; Apheresis Related Complication
Keywords: Apheresis; DFPP; ANCA associated vasculitis; Goodpasture syndrome; Arterio veinous fistula; Arterio veinous graft
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Anti-Glomerular Basement Membrane Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to describe vascular access complications which are used for therapeutic apheresis in Nephrology.

DETAILED DESCRIPTION:
The aim of this study is to describe vascular access complications which are used for therapeutic apheresis in Nephrology.

Complications may include arterio-veinous fistula or graft (AVF or AVG) thrombosis with or without known stenosis; AVF or AVG or central veinous catheter (CVC) infections and CVC dysfunctions.

The investigators may enroll all patients receveing therapeutic apheresis for nephrologic indications in North East France.

Nephrologics indications include :

* acute or active antibody mediated rejection (ABMR),
* Goodpasture disease,
* ANCA vasculitis,
* thrombotic microangiopathy (TMA),
* Focal segmental glomerulosclerosis (FSGS),
* HLA or ABO desensitization for kidney transplantation.

Data inclusion period is from June 2020 to June 2022.

The aim of the study is to describe the proportion and type of complication in the population of patient receving therapeutic apheresis for nephrologic disease in the North East France. Te investigators will study the risk factors that are associated with this complications.

The second aim of the study is to describe the population of patient receving therapeutic apheresis in our unit and in our region.

ELIGIBILITY:
Inclusion Criteria:

* patients in nephrology receiveing apheresis treatment by filtration or double filtration

Exclusion Criteria:

* apheresis treatment for other indications
* centrifugation apheresis treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients in nephrology receiveing apheresis treatment by filtration or double filtration with arterioveinous fistula or arterioveinous graft or central veinous catheter
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Vascular access Complication (catheter or AVF/AVG thrombosis/infection) rate in therapeutic apheresis among nephrological diseases | june 2020 june 2022
  Percent of patient with Vascular access Complication

SECONDARY OUTCOMES:
Description of population enrolled | june 2020 june 2022
  Description of population treated by therapeutic apheresis in Northeast France
Comparison of complications rate with literature datas | june 2020 june 2022

CONTACTS AND LOCATIONS:
Overall Officials: Luc Frimat, MD PhD, Principal Investigator — CHRU NANCY DRCI
Locations (1):
- Central Hospital, Nancy, France

IPD SHARING:
Plan to Share IPD: No